CLINICAL TRIAL: NCT00810342
Title: Physical Activity in Women With Infants
Acronym: "NaMikimiki"
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CA115614; 5R01CA115614 (NIH); R01CA115614-03S1 (NIH)
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Results first posted 2015-06-04 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-01

CONDITIONS: Physical Activity
Keywords: physical activity standard; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1- physical activity tailored (Experimental): Tailored telephone counseling about how to become more physically active and goal setting. Email feedback on physical activity progress. Website listing resources new mothers can use to become more active.
  Interventions: Behavioral: physical activity tailored
- 2 - physical activity standard (Active Comparator): Standard Website resources / information on physical activity
  Interventions: Behavioral: physical activity standard

INTERVENTIONS:
Behavioral: physical activity tailored — tailored telephone counseling, email feedback, and website resources over 12 months
  Other Names: tailored exercise advice
  Arms: 1- physical activity tailored
Behavioral: physical activity standard — standard print and website information on how to become more active
  Other Names: standard information about physical activity
  Arms: 2 - physical activity standard

SUMMARY:
This is a study testing ways to motivate new mothers to become more physically active over a one year period.

DETAILED DESCRIPTION:
Mothers of an infant are much less likely to exercise regularly compared with women who have older children or no children. This low level of physical activity (PA) contributes to postpartum weight retention which can predict levels of obesity up to 15 years later. Ethnic minorities have higher rates of inactivity and gain more weight following childbirth, which places them at increased risk for cancer and other chronic diseases consistent with known health disparities for these ethnic groups. Few PA interventions have been designed to increase PA in women with an infant, especially ethnic minority women. This study will test the efficacy of a tailored intervention to increase and maintain PA in a multiethnic population of 268 young, healthy postpartum women living in Hawaii. Women will be recruited from health care settings, mother/baby support groups, and from the media campaigns(TV, radio, newspaper, parents magazines). Subjects will be randomly assigned to either a tailored postpartum counseling intervention on PA or standard care for PA. The tailored PA intervention will address key personal, social, and environmental factors derived from Social Cognitive Theory and the Transtheoretical Model. Also, multimodal contacts (telephone, e-mail, website) will be used to deliver theoretically-derived, culturally sensitive PA counseling,behavioral skills training (e.g., goal setting), and local resources/referrals tailored to a mother with an infant. The standard care condition receives American Heart Association/American College of Sports Medicine print materials/e-mails and referral to PA internet resources.

The primary PA outcome is minutes of moderate/vigorous physical activity (MVPA) per week, as measured by the Active Australia Questionnaire, with validation by accelerometers worn by all subjects. Condition differences in the initiation of PA will be tested at 6 and 12 months post-baseline. Key psychosocial, physiological, and cultural factors will be tested as mediators or moderators of PA, for example: self-efficacy, social support, processes of change, ethnicity, BMI, and cultural values. This study will serve as a model for the design and implementation of PA interventions for at-risk ethnic minority postpartum women.

ELIGIBILITY:
Inclusion Criteria:

* mother of infant aged 2-12 months
* sedentary
* healthy, able to do moderate intensity physical activity
* BMI = 18.5-40
* not planning to become pregnant in next year
* woman aged 18-45
* able speak and read English

Exclusion Criteria:

* pregnant
* planning to leave Oahu, Hawaii in the next year (permanently move away)
* a diagnosis of cancer, coronary heart disease (including atrial fibrillation), insulin-dependent diabetes mellitus (IDDM), and other atherosclerotic cardiovascular diseases (e.g., stroke),

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 311 (Actual)
Dates: Start 2008-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl L Albright, PhD, MPH, Principal Investigator — University of Hawaii, School of Nursing and Dental Hygiene
Locations (1):
- University of Hawaii School of Nursing, Honolulu, Hawaii, United States

REFERENCES:
- [Derived] Albright CL, Saiki K, Steffen AD, Woekel E. What barriers thwart postpartum women's physical activity goals during a 12-month intervention? A process evaluation of the Na Mikimiki Project. Women Health. 2015;55(1):1-21. doi: 10.1080/03630242.2014.972014. Epub 2015 Jan 30. PMID 25402618
- [Derived] Albright CL, Steffen AD, Novotny R, Nigg CR, Wilkens LR, Saiki K, Yamada P, Hedemark B, Maddock JE, Dunn AL, Brown WJ. Baseline results from Hawaii's Na Mikimiki Project: a physical activity intervention tailored to multiethnic postpartum women. Women Health. 2012;52(3):265-91. doi: 10.1080/03630242.2012.662935. PMID 22533900

RESULTS

PARTICIPANT FLOW:
Groups:
- 1- Tailored: Tailored telephone counseling about how to become more physically active. Email feedback on physical activity progress. Website listing resources new mothers can use to become more active.
  physical activity tailored: tailored telephone counseling, email feedback, and website resources over 12 months
- 2 - Standard: Website resources on physical activity
  physical activity: standard print and website information on how to become more active
Period: Month 1 Follow-up
Arm/Group | 1- Tailored | 2 - Standard
Started | 154 | 157
Completed | 149 | 155
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 4 | 2
Not completed — Pregnancy | 1 | 0
Period: 6-month Follow-up
Arm/Group | 1- Tailored | 2 - Standard
Started | 149 | 155
Completed | 125 | 147
Not Completed | 24 | 8
Not completed — Lost to Follow-up | 18 | 6
Not completed — Pregnancy | 6 | 2
Period: 12-month Followup
Arm/Group | 1- Tailored | 2 - Standard
Started | 125 | 147
Completed | 113 | 136
Not Completed | 12 | 11
Not completed — Pregnancy | 9 | 10
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Population: Chi square test for differences in proportions; t test for differences in means
Groups:
- Total: Total of all reporting groups
Arm/Group | 1- Tailored | 2 - Standard | Total
Number analyzed (Participants) | 154 | 157 | 311
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (5.5) | 32.1 (5.9) | 31.8 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 157 | 311
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 30 | 54
  Not Hispanic or Latino | 128 | 124 | 252
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 53 | 52 | 105
  Native Hawaiian or Other Pacific Islander | 49 | 49 | 98
  Black or African American | 4 | 4 | 8
  White | 20 | 27 | 47
  More than one race | 27 | 24 | 51
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 154 | 157 | 311
Minutes per week of moderate-to-vigorous physical activity [Mean (Inter-Quartile Range); unit: minutes per week] | 44 [41 to 47] | 46 [42 to 49] | 45 [41.5 to 48]

OUTCOME MEASURES:

1. Primary Outcome: Minutes of Moderate or Vigorous Physical Activity Per Week After 12-months
Description: Self reported minutes of moderate or vigorous physical activity per week after 12-months
Time Frame: 12 months
Population: Treatment effect was assessed by a mixed growth model and the F test of the fixed 2-way interaction parameter for time and study condition for overall and of the 3-way interaction parameter for characteristic level, time, and study condition. Adjusted for age, race, BMI, education, #children, employment, depression, baby's age, years in Hawaii
Measure: Mean (Inter-Quartile Range); unit: minutes per week moderate-to-vigorous PA
Arm/Group | 1- Tailored | 2 - Standard
Number analyzed (Participants) | 113 | 136
minutes per week moderate-to-vigorous PA | 246 [222 to 272] | 156 [140 to 173]

2. Secondary Outcome: Accelerometer Collected Moderate to Vigorous Physical Activity
Description: Participant's physical activity (overall moderate-to-vigorous physical activity above 2.9 metabolic equivalents (METs) collected via an accelerometer over 12 months
Time Frame: 12-Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: minutes per week moderate-to-vigorous PA
Arm/Group | 1- Physical Activity Tailored | 2 - Physical Activity Standard
Number analyzed (Participants) | 113 | 136
minutes per week moderate-to-vigorous PA | 215 [200 to 229] | 203 [189 to 217]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | 1- Tailored | 2 - Standard
Serious Adverse Events (participants affected / at risk) | 2/154 | 2/157
Other Adverse Events (participants affected / at risk) | 4/154 | 2/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1- Tailored (N=154) | 2 - Standard (N=157)
Intracranial tumor (disorder) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (disorder) Blackout (disorder) Spinal cord injury (disorder) (Nervous system disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1- Tailored (N=154) | 2 - Standard (N=157)
Fracture elbow (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
suicidal thoughts (finding) (Psychiatric disorders) | 1 (1) | 0 (0)
Fracture ribs (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fracture - Toe (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No